CLINICAL TRIAL: NCT06273787
Title: Effect of Diaphragmatic Release in Sleep Quality During Pregnancy, Randomized Controlled Trail
Brief Title: Effect of Diaphragmatic Release in Sleep Quality During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, shaimaa Mohamed hamed, Lecturer of physical therapy for women's health in MTIU, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mitu
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: SLEEP APNEA PREGNANCY

STUDY DESIGN:
Intervention Model Description: Parallel Assignment group a : Diaphragmatic Release in addition to positioning instruction group b: positioning instruction
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diaphragmatic release (Experimental): diaphragmatic myofascial release
  Interventions: Other: diaphragmatic release
- positioning (Active Comparator): positioning instruction for sleep apnea
  Interventions: Other: diaphragmatic release

INTERVENTIONS:
Other: diaphragmatic release — diaphragmatic myofascial release for 1 months 3 sessions per week

SUMMARY:
Sleep disordered breathing (SDB) is very common during pregnancy, and is most likely explained by hormonal, physiological and physical changes. Maternal obesity, one of the major risk factors for SDB, together with physiological changes in pregnancy may predispose women to develop SDB. SDB has been associated with poor maternal and fetal outcomes. Thus, early identification, diagnosis and treatment of SDB are important in pregnancy.

DETAILED DESCRIPTION:
The present study will be conducted to add a new information to the body of knowledge of physical therapy profession as it will provide scientific basis for the clinical application of diaphragmatic release in sleep disordered breathing during pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (at third trimester), diagnosed with sleep disordered breathing by the gynaecologist.
* Their ages will range from 30- 40 years old .
* Their BMI will be 25 to 30kg/m2.
* All are multipara.

Exclusion criteria:

Women will be excluded from the study if they have:

* Previous pulmonary surgery.
* any pulmonary diseases.
* Asthma.
* Neurological disorders
* Musculoskeletal disorders (severe osteoarthritis, osteoporosis)

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant female
Enrollment: 44 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-03-17 (Estimated)

PRIMARY OUTCOMES:
pittshurgh sleep quality index | 1 month
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Developed by researchers at the University of Pittsburgh,

SECONDARY OUTCOMES:
diaphragmatic excursion assessment | 1 month
  diaphragmatic excursion assessment is that measures the movement of the thoracic diaphragm during breathing. Normal diaphragmatic excursion should be 3-5 cm, but can be increased in well-conditioned persons to 7-8 cm2.

CONTACTS AND LOCATIONS:
Locations (1):
- MTI, Cairo, Egypt